CLINICAL TRIAL: NCT02148536
Title: Effect of Transjugular Intrahepatic Portosystemic Shunt on Oxygenation in Cirrhotic Patients With Hepatopulmonary Syndrome
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li, Professor, West China Hospital
Other Study IDs: WCH-2014-034
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hepatopulmonary Syndrome
MeSH Terms: conditions — Hepatopulmonary Syndrome | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — aterial and venous blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HPS-TIPS group
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt

SUMMARY:
To prospectively investigate the effect of transjugular intrahepatic portosystemic shunt (TIPS) on oxygenation in cirrhotic patients with hepatopulmonary syndrome (HPS).

ELIGIBILITY:
Inclusion Criteria:

* Presence of cirrhosis
* Alveolar-arterial oxygen gradient ≥ 15 mm Hg (≥ 20 mm Hg for age > 64 years)
* Positive contrast-enhanced echocardiography

Exclusion Criteria:

* Age of less than 18 years
* Intrinsic cardiopulmonary disease
* Malignancy
* Active infection
* Pregnancy
* Previous shunt therapy
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients with hepatopulmonary syndrome undergoing transjugular intrahepatic portosystemic shunt for any indication at West China Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Alveolar-arterial oxygen gradient (PA-a,O2) | 12 Weeks

SECONDARY OUTCOMES:
Macroaggregated albumin (MAA) shunt fraction | 12 Weeks
Exhaled nitric oxide (eNO) | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan university, Chengdu, Sichuan, China